CLINICAL TRIAL: NCT05261165
Title: Effect of a Uterine Manipulator on the Incidence of Lymphovascular Propagation (LVSI) in Treatment of Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other)
Responsible Party: Principal Investigator, Boris Hudec, MD, Mr., F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica
Other Study IDs: 29/2021
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Endometrial Cancer; LVSI
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NonManip: In the group of female patients operated without a uterine manipulator (NonManip), we included the female patients who were operated by abdominal approach without no need to use a manipulator. These female patients did not meet the predominantly anesthesiological requirements for the tolerance of the Trendelenburg position; respectively, the likelihood of adhesions in the abdominal cavity after previous laparotomy operations was there. Therefore, from a safety point of view, due to the risk of damage to the abdominal organs and the need for extensive adhesiolysis, the primary endoscopic surgery was not performed.
  Interventions: Procedure: hysterectomy
- Manip: The female patients suitable for endoscopic performance to laparoscopic, respectively the robotic hysterectomies, in whom the use of a uterine manipulator (Manip) was planned, were assigned random into two groups.
  Interventions: Procedure: hysterectomy
- ManipHe: Subgroup of Manip group patients, in whome we used the Hegar's dilator as intrauterine manipulator.
  Interventions: Procedure: hysterectomy
- ManipKoRu: Subgroup of Manip group patients, in whome we used the Koh-Rumi device as intrauterine manipulator.
  Interventions: Procedure: hysterectomy

INTERVENTIONS:
Procedure: hysterectomy — Hysterectomy as primary surgical treatment of endometrial cancer. Abdominal laparotomy approach was performed without intrauterine manipulator (NonManip). Endoscopic - total laparoscopic hysterectomy, laparoscopic assisted vaginal hysterectomy or robotic hysterectomy was performed with use of intrauterine manipulator (Manip). It was Hegar dilatator (ManipHe) or Koh-Rumi device (ManipKoRu).

SUMMARY:
We retrospectively analyzed data and compared the impact of intrauterine manipulators on incidence of LVSI in endometrial cancer patients treated at our department.

DETAILED DESCRIPTION:
Endometrial cancers are among the epithelial malignancies of the lining in the uterine cavity. Standard treatment is surgical, which includes a hysterectomy. The invasion of carcinoma into the lymphovascular space (LVSI - lymphovascular space invasion) is considered a risk factor for the course of the disease Based on the recommended procedures of ESGO-ESTRO-ESP (2020) in the management of endometrial cancer, in the event of significant LVSI positivity, the female patients are included in the upper-medium risk group. A confirmation of LVSI in the preparation is of diagnostic, therapeutic and theoretical importance. During endoscopy approach, we use two types of uterine manipulators, namely the Koh-RUMI manipulator (Cooper Surgical) and the Hegar dilatator along with the McCartney tube (LiNA Medical). We analyzed data and compared the impact of intrauterine manipulators on the incidence of LVSI. In addition, we analyzed tumor grading, invasion and primary histology obtaining methods - curettage or hysteroscopy in correlation to incidence of LVSI.

ELIGIBILITY:
Inclusion Criteria:

* endometrioid endometrial cancer,
* planned primary surgical treatment - hysterectomy,
* medical condition enabling anesthesia and surgery,
* pre-surgical clinically-determined affecting of the uterine according to MRI or ultrasound - cT1a or cT1b

Exclusion Criteria:

* non-endometrioid type of tumor in definitive histology,
* stage 2 of a disease and higher,
* previous chemo or radiotherapy,
* inability to adequately complete the surgery,
* uterine perforation during surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women diagnosed with endometrial cancer, planned to primary surgical treatment - hysterectomy.
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
LVSI and intrauterine manipulator | oct. 2015 - jan. 2021
  Finding of the difference in the incidence of LVSI in female patients with and without an intrauterine manipulator

SECONDARY OUTCOMES:
LVSI and type of intrauterine manipulator | oct. 2015 - jan. 2021
  The effect of a type of an intrauterine manipulator on the incidence of LVSI

OTHER OUTCOMES:
LVSI and grading of tumor | oct. 2015 - jan. 2021
  Connection between grading of tumor and incidence of LVSI
LVSI and myometrial invasion | oct. 2015 - jan. 2021
  Connection between myometrial invasion of tumor and incidence of LVSI
LVSI and primary histology procedure | oct. 2015 - jan. 2021
  Method of obtaining primary histology, hysteroscopy or curettage in connection to incidence of LVSI.

CONTACTS AND LOCATIONS:
Locations (1):
- F.D. Roosevelt Teaching Hospital with Policlinic, Banská Bystrica, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hudec B, Dokus K, Urdzik P, Skolka R, Konarcikova T, Smitka M. Influence of uterine manipulator use on the incidence of lymphovascular propagation in the treatment of endometrial cancer. Minim Invasive Ther Allied Technol. 2023 Feb;32(1):12-17. doi: 10.1080/13645706.2022.2153342. Epub 2022 Dec 21. PMID 36542513